CLINICAL TRIAL: NCT01211093
Title: The Acute Effects of Whole Body Vibration Training With Different Frequencies on Neuromotor Performance in Individuals With Stroke
Brief Title: Acute Effects of Whole Body Vibration in Chronic Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Marco Yiu-Chung Pang, Associate Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: HSEARS20091016003-01
Record Dates: First submitted 2010-09-17; First posted 2010-09-29 (Estimated); Last update posted 2012-11-28 (Estimated); Status verified 2012-11

CONDITIONS: Stroke
Keywords: vibration; muscle; cerebrovascular accident; exercise; rehabilitation
MeSH Terms: conditions — Stroke; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- High frequency whole body vibration (Experimental): This group will receive a single 10-minute session of WBV therapy. The frequency of the vibration signals will be set at 30Hz.
  Interventions: Procedure: High frequency whole body vibration
- low frequency whole body vibration (Active Comparator): This group will receive a single 10-minute session of WBV. The frequency of the vibration signals will be set at 20 Hz.
  Interventions: Procedure: Low frequency whole body vibration
- Control (Active Comparator): This group will stand on the same vibration platform for 10 minutes, but no vibration will be given.
  Interventions: Procedure: control

INTERVENTIONS:
Procedure: High frequency whole body vibration — 1 single session (10 minutes) of whole body vibration therapy at 30 Hz
  Other Names: Whole body vibration therapy (30Hz)
  Arms: High frequency whole body vibration
Procedure: Low frequency whole body vibration — 1 single session of whole body vibration therapy at 20 Hz
  Other Names: Whole body vibration therapy (20Hz)
  Arms: low frequency whole body vibration
Procedure: control — 1 single session of standing on the vibration platform, with no vibration signals delivered.
  Arms: Control

SUMMARY:
Whole body vibration has been found to be useful in promoting bone health, balance, and muscle performance in older adults. The overall aim of the proposed study is to determine whether whole body vibration (WBV) has immediate beneficial effect in neuromotor performance in patients with stroke. It is hypothesized that a single session of WBV will induce significant improvement in leg muscle strength in people with chronic stroke.

ELIGIBILITY:
Inclusion Criteria:

* a diagnosis of stroke
* stroke onset >6 months
* >18 years of age
* >able to walk for short distance independently with or without walking aid
* able to understand simple verbal commands

Exclusion Criteria:

* other neurological conditions
* peripheral vascular disease
* vestibular disorders
* significant musculoskeletal disorders (e.g. rheumatoid arthritis)
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2009-11; Primary Completion 2013-04 (Estimated); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
knee extension isokinetic strength | 2 weeks

SECONDARY OUTCOMES:
Muscle activity (electromyography) of knee extensors | during treatment
knee extension isometric strength | 2 weeks
knee flexion isometric strength | 2 weeks
knee flexion isokinetic strength | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Marco YC Pang, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, China